CLINICAL TRIAL: NCT02637700
Title: Intravenous Immunoglobulin Therapy for Small Fiber Neuropathy: a Randomized, Double-blind, Placebo-controlled Study on Efficacy and Safety.
Brief Title: Intravenous Immunoglobulin Therapy for Small Fiber Neuropathy
Acronym: IVIg-SFN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Catharina G. Faber, MD, PhD, Academisch Ziekenhuis Maastricht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVIg-SFN; 2015-002624-31 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Small Fiber Neuropathy
Keywords: Small Fiber Neuropathy; Painful Neuropathy; Intravenous Immunoglobulin Therapy
MeSH Terms: conditions — Small Fiber Neuropathy; Neuropathy, Painful | interventions — Immunoglobulins, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Immunoglobulin (Experimental): Patients with skin biopsy proven idiopathic Small Fiber Neuropathy in this arm will receive intravenous immunoglobulin.
  Interventions: Drug: Intravenous Immunoglobulin
- Placebo (Saline 0.9%) (Placebo Comparator): Patients with skin biopsy proven idiopathic Small Fiber Neuropathy in this arm will receive placebo (saline 0.9%).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous Immunoglobulin — Comparison between intravenous immunoglobulin and placebo (saline 0.9%).
  Other Names: Gamunex
  Arms: Intravenous Immunoglobulin
Drug: Placebo — Comparison between placebo (saline 0.9%) and intravenous immunoglobulin.
  Other Names: Saline (0.9%)
  Arms: Placebo (Saline 0.9%)

SUMMARY:
Small fiber neuropathy (SFN) is the most common cause of neuropathic pain in peripheral neuropathies, with a prevalence of at least 53/100.000. Patients with SFN may have excruciating pain and current anti-neuropathic and other pain drugs do not relief pain substantially.

Several studies suggested an immunological basis in SFN and case studies have reported efficacy of treatment with intravenous immunoglobulin (IVIg) in patients with SFN. It is therefore conceivable that immunological mechanisms play a role in idiopathic SFN (I-SFN). However, to date no randomized controlled study with IVIg in patients with SFN has been performed. The aim of the current study is to investigate the efficacy and safety of IVIg in patients with I-SFN in a randomized, double-blind, placebo-controlled study.

The objective of the study is to evaluate the efficacy of IVIg treatment (4 courses of treatment, 3 weeks apart) compared to placebo on pain alleviation.

DETAILED DESCRIPTION:
Small nerve fiber neuropathy (SFN) is a disorder of thinly myelinated and unmyelinated nerve fibers recently recognized as a distinct clinical syndrome, with a minimum incidence of 12 per 100.000 and a minimum prevalence of 53 per 100.000. The clinical picture is typically dominated by neuropathic pain, often with a burning quality, and autonomic symptoms. The diagnosis of SFN is usually made on the basis of the clinical picture, no involvement of large nerve fibers at neurological examination and normal nerve conduction studies (NCS), and is confirmed by demonstration of reduced intra-epidermal nerve fiber density (IENFD) or abnormal quantitative sensory testing (QST). Despite intensive search for underlying causes such as diabetes mellitus, impaired glucose tolerance, Fabry's disease, hereditary disorders, celiac disease, sarcoidosis, HIV and other systemic illnesses which may be potentially treatable, the proportion of patients with idiopathic SFN (I-SFN) remains substantial, ranging in different series from 24% up to 93%. It is conceivable that immunological mechanisms play a role in patients with I-SFN, since several immune-mediated diseases, such as sarcoidosis, Sjogren's disease and systemic lupus erythematosis may cause SFN. Auto-antibodies have also been reported in patients with SFN. Moreover, inflammatory changes in nerves have been found. Elevated pro-inflammatory cytokines have been suggested to be involved in the pathophysiology of pain in SFN.

In other immune-mediated neuropathies, such as chronic inflammatory demyelinating polyneuropathy, treatment with intravenous immunoglobulin (IVIg) has proven to be efficacious. Moreover, some case studies in patients with SFN and chronic pain have also reported effect of immunomodulating therapy. Pain reduction with IVIg treatment has also been summarized recently.

Intravenous infusion of high doses of pooled immunoglobulin G (IgG) molecules from thousands of donors (IVIg therapy) represents an efficient anti-inflammatory treatment for many autoimmune diseases. Paradoxically, IgG can exert both pro- and anti-inflammatory activities, depending upon its concentration. When administered in high concentrations, IVIg has anti-inflammatory properties. How this anti-inflammatory effect is mediated has not yet been fully elucidated. Several mutually nonexclusive mechanisms have been proposed, including modulation of the expression and function of the Fc fragment of IgG to IgG-specific receptors, interference with activation of the complement cascade and the cytokine network, neutralization of autoantibodies and regulation of cell proliferation. However, the exact mechanism of IVIg in the treatment of inflammatory neuropathies has not been elucidated.

Side effects of IVIg treatment are usually transient (chills, headache, dizziness, fever, vomiting, nausea, arthralgia, low blood pressure and moderate low back pain may occur occasionally).

Sudden fall in blood pressure and anaphylactic shock are rare. More severe side effect are extremely rare (reversible aseptic meningitis, transient cutaneous reactions, reversible haemolytic reactions, haemolytic anemia, and thromboembolic events).

SFN is considered the most common cause of neuropathic pain in peripheral neuropathies. Patients with SFN have reported having excruciating pain, since current anti-neuropathic and other pain drugs do not relief pain substantially. SFN interferes with daily functioning and may lead to a decrement in quality of life expectations. Therefore, a better treatment is warranted. The aim of the current pilot study is to investigate the efficacy and safety of IVIg in patients with I-SFN in a randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Patients can only participate when they are living in the Netherlands.

Inclusion Criteria:

* 18 years or older.
* Skin-biopsy proven idiopathic SFN or idiopathic painful neuropathy with predominantly SFN pattern
* Pain intensity rated ≥ 5 on the PI-NRS (maximum pain) or on the neuropathic pain scale,36,37 question number 1 for at least 12 weeks before the study as declared by each patient to the best of their knowledge; if available, medical records of each patient will be consulted on the reported pain intensity.
* Each subject will receive an information leaflet and an informed consent form. Subjects must give informed consent by signing and dating prior to study entry.
* Eligible patients must be willing to complete all study-related activities and examination required by the protocol (see Tables 1-4).

Exclusion Criteria:

* Are unable or unwilling to provide written informed consent.
* Have predominant clinical picture of large nerve fiber involvement (i.e., weakness, loss of vibration sense, hypo-/areflexia).
* Had treatment with IVIg or any other immunomodulatory/immunosuppressive agents (e.g., steroids) within the last 12 weeks prior to the date of informed consent.
* Have an underlying cause of SFN (diabetes, SCN9A/10A/11A mutations, hypothyroidism, renal failure, vitamin B12 deficiency, monoclonal gammopathy, alcohol abuse (more than 5 IU/day), malignancies, drugs that cause neuropathy (e.g. chemotherapy, amiodarone, propafenone)).
* Have a history of anaphylaxis or severe systemic response to immunoglobulin or with a blood product.
* Have cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease, or history of congestive heart failure, severe hypertension (diastolic blood pressure >120 mmHg or systolic >170 mmHg).
* Are females who are pregnant, breast-feeding, or if of childbearing potential, or unwilling to practice adequate contraception throughout the study.
* Have known hyperviscosity.
* Have a history of renal insufficiency or high serum creatinine levels (MDRD <30).
* Have known selective immunoglobulin A (IgA) deficiency.
* Have conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
* Have a known hypercoagulable state.
* Are mentally challenged adult subjects unable to give independent informed consent.
* The use of pain (analgesic/anti-neuropathic) medication is allowed, but only if dosages are remained unchanged for at least 30 days prior to randomization. A change in dosage of these drugs will not be allowed throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Numerical Rating Scale (PI-NRS) | Mean weekly pain intensity is assessed twice a week for a period of three months

SECONDARY OUTCOMES:
Change in Pain Intensity Numerical Ratings Scale (PI-NRS) | The nocturnal pain intensity will be assessed twice a week for a period of three months
Patient Global Impression of Change (PGIC) | The global impression of change will be measured 5 times in three months
Change in Small Fiber Neuropathy Symptoms Inventory Questionnaire (SFN-SIQ) | This will be measured 5 times in three months
Change in Neuropathic Pain Scale (NPS) | This will be measured 5 times in three months
Change in Small Fiber Neuropathy Rasch-Built Overall Disability Scale (SFN-RODS) | This will be measured 5 times in three months
Pain relief questionnaire | This will be measured 5 times in three months
Change in Daily sleep interference scale (DSIS) | This will be measured 5 times in three months
Change in SF-36 | This will be measured 5 times in three months
Adverse events, laboratory safety tests, vital signs. | This will be measured 8 times in three months

CONTACTS AND LOCATIONS:
Overall Officials: Catharina G Faber, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Geerts M, de Greef BTA, Sopacua M, van Kuijk SMJ, Hoeijmakers JGJ, Faber CG, Merkies ISJ. Intravenous Immunoglobulin Therapy in Patients With Painful Idiopathic Small Fiber Neuropathy. Neurology. 2021 May 18;96(20):e2534-e2545. doi: 10.1212/WNL.0000000000011919. Epub 2021 Mar 25. PMID 33766992
- [Derived] de Greef BT, Geerts M, Hoeijmakers JG, Faber CG, Merkies IS. Intravenous immunoglobulin therapy for small fiber neuropathy: study protocol for a randomized controlled trial. Trials. 2016 Jul 20;17(1):330. doi: 10.1186/s13063-016-1450-x. PMID 27439408